CLINICAL TRIAL: NCT02816840
Title: Pilot Study of the Incorporation of PET-CT/MRI in the Radiotherapy for Prostate Cancer
Brief Title: PET-CT/MRI in the Radiotherapy for Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Longzhen Zhang, professor, Xuzhou Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL015-01
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radiotherapy; PET-CT/MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PET-CT (Experimental): Patients in this arm take radiotherapy positioning with PET-CT.
  Interventions: Radiation: PET-CT
- PET-MRI (Experimental): Patients in this arm take radiotherapy positioning with PET-MRI.
  Interventions: Radiation: PET-MRI
- Computed Tomography (No Intervention): Patients in this arm take radiotherapy positioning with CT.

INTERVENTIONS:
Radiation: PET-CT — Patients in this arm take radiotherapy positioning with PET-CT.
  Arms: PET-CT
Radiation: PET-MRI — Patients in this arm take radiotherapy positioning with PET-MRI.
  Arms: PET-MRI

SUMMARY:
The trial is to explore new and effective techniques in the treatment of prostate cancer and evaluate the role of PET-CT / MRI played in radiotherapy. Intensity modulated radiation therapy(IMRT) is adopted with all patients and the efficacy assessment for the prostate cancer will be examined with PET / CT or CT in three months after radiotherapy.

DETAILED DESCRIPTION:
All participants judged to have prostate cancer with stage Ⅲ-Ⅳand considered able to conduct radiotherapy. 180 patients will be enrolled in the trial and randomly divided into three groups. Three arms are respectively treated with CT、18F-FDG PET/CT、18F-FDG PET/MRI. The images were passed in three-dimensional treatment planning system, using software manually fusion and reconstruction of PET and CT. All patients adopt IMRT for the radiotherapy with 70Gy-80Gy. Three months after radiotherapy, solid tumer size for the prostate cancer will be assesed with PET / CT or CT. Early radiation reactions are evaluated by the United States RTOG (RTOG) acute response evaluation criteria, and late radiation reaction are evaluated with RTOG and the European Radiation Therapy Oncology Organization (EORTC). Before and after radiotherapy treatment,the tumor-associated marker of PSA will be monitored and the patients are regularly followed-up in the next three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed prostate cancer
* Staged with Ⅲ-Ⅳ prostate cancer
* Aged from 18 to 65 years old
* Quality of life score (Karnofsky performance score) > 70
* No distant metastasis
* No serious internal diseases may affect the treatment plan
* No previous history of prostate radiation therapy
* Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Distant metastasis
* Accompanied by other malignancies
* Previous history of prostate radiation therapy
* Pregnant or lactating women
* History of allergic reaction to iodinated, non-iodinated, and/or gadolinium contrast agents
* Liver and kidney dysfunction
* Pacemaker or other metallic devices that would prevent MRI imaging from being performed
* Patients quit during the treatment or violate of the study protocol caused by other factors
* Any reason that, in the option of the investigator, contraindicates that the patient participates in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Solid tumor size | Three months
  Three months after radiotherapy, the efficacy assessment for the prostate cancer will be examined with PET/CT or CT.

SECONDARY OUTCOMES:
Relapse-free survival | Three years

OTHER OUTCOMES:
Overall survival | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Longzhen Zhang, MD, Principal Investigator — Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: No